CLINICAL TRIAL: NCT00533156
Title: Feasibility Study of the 7F Ensure Medical Plug Arterial Closure System (PACS, 7F)
Brief Title: Plug Arterial Closure System (PACS, 7F)
Acronym: PACS 7F
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Collaborators: Ensure Medical (Industry)
Responsible Party: Chao-Chin Chen, Vice President, Ensure Medical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMI 07-02
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Angioplasty, Transluminal, Percutaneous Coronary; Coronary Arteriosclerosis
Keywords: Closure Device; Angiography; Angioplasty; Hemostasis; Heart Catheterization; Vascular Closure; Peripheral Closure; Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vascular access site closure (7F Ensure)

SUMMARY:
The purpose of this study is to assess the safety and feasibility of the 7F Ensure Medical Vascular Closure Devices to facilitate hemostasis in patients undergoing diagnostic or interventional coronary procedures using a standard 7F introducer sheath.

DETAILED DESCRIPTION:
Achieving hemostasis at the arterial puncture site after percutaneous cardiac catheterization is a potential cause of bleeding, hematomas, pseudoaneurysms, and various other vascular complications. Hemostasis at the femoral artery access site after diagnostic or interventional procedures is typically achieved using either manual compression or the deployment of a vascular closure device. Manual compression is time consuming for the health-care provider, and painful for the patient. In addition, prolonged periods of immobilization and bed rest may be required. Vascular closure devices have been developed to avoid manual compression, shorten bed rest, and allow earlier ambulation.

The Ensure Medical Vascular Closure device (VCD) is intended for femoral artery puncture site closure in patients who have undergone coronary catheterizations using a standard 7F introducer sheath. The device is comprised of a bio-absorbable plug and a plug delivery system. The plug delivery system is designed to position the bio-absorbable plug to the extravascular surface of the femoral artery access site, facilitating a hemostasis response. The Ensure Medical VCD has been studied in a prior feasibility trial of 149 patients utilizing a 6F introducer sheath, which demonstrated that: (1) the device could be used to successfully obtain rapid hemostasis and early ambulation in patients undergoing catheterization procedures; and (2) the low incidence and relatively minor nature of the observed closure related complications suggests that the device is safe for its intended purpose.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a coronary diagnostic or interventional procedure
* Able to undergo emergent vascular surgery if a complication requires it
* 7F arterial puncture located in the common femoral artery
* Femoral artery has a lumen diameter of at least 5 mm

Exclusion Criteria:

* Arterial puncture in the femoral artery of both legs
* Prior target artery closure with any vascular closure device, or closure with manual compression within 30 days prior to catheterization
* Patients who bruise or bleed easily or with a history of significant bleeding or platelet disorders
* Acute ST-elevation myocardial infarction within 48 hours prior to catheterization
* Uncontrolled hypertension at time of vessel closure
* Elevated Activated Clotting Time at time of vessel closure
* Ineligible for in-catheterization lab introducer sheath removal
* Concurrent participation in another investigational device or drug trial
* Thrombolytic therapy, bivalirudin, other thrombin-specific anticoagulants, or low molecular weight heparin within 24 hours prior to catheterization
* Preexisting hematoma, arteriovenous fistula, or pseudoaneurysm at the vessel access site prior to femoral artery closure
* Prior femoral vascular surgery or vascular graft in region of access site
* Femoral artery is tortuous or requires an introducer sheath longer than 11 cm
* Fluoroscopically visible calcium, atherosclerotic disease, or stent within 1 cm of the puncture site that would interfere with the operation of the experimental device
* Difficulty in obtaining vascular access resulting in multiple arterial punctures and/or posterior arterial puncture
* Antegrade vascular puncture
* Body Mass Index over 40 kg/m2
* Symptomatic leg ischemia in the target limb including severe claudication or weak/absent pulse
* Femoral artery diameter stenosis exceeding 50%
* Pre-existing severe non-cardiac systemic disease or terminal illness
* Planned arterial access at the same access site within 30 days of catheterization
* Extended hospitalization (e.g. CABG surgery)
* Pre-existing systemic or cutaneous infection
* Prior use of an intra-aortic balloon pump through the arterial access site
* Cardiogenic shock during or immediately following the catheterization
* Patient is unable to ambulate at baseline
* Patient is known or suspected to be pregnant or is lactating
* Patient is unavailable for follow-up
* Any angiographic or clinical evidence that the physician feels would place the patient at increased risk with the use of the experimental device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to hemostasis following vessel access site closure | 5 minutes post procedure
Time to ambulation following vessel access site closure | Post-procedure
Combined rate of closure related major adverse events at 30 days | Through 30 days

SECONDARY OUTCOMES:
Device success (initial hemostasis within 5 minutes) | Within 5 minutes
Procedural success on day of catheterization and at 30 days (initial hemostasis by non-randomized treatment without closure related serious adverse events) | Through 30 days
Time patient is deemed eligible for hospital discharge relative to their access site closure | Up to hospital discharge
Time patient is discharged from the hospital | Patient discharge
Known events associated with vascular closure devices | Through 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Luna, MD, Principal Investigator — HOSPITAL ALMATER
Locations (1):
- Hospital Almater, Mexicali, Estado de Baja California, Mexico